CLINICAL TRIAL: NCT07059351
Title: Oral Status as Predictors of Stroke-Associated Pneumonia and Swallowing Recovery in Patients With Post-Stroke Dysphagia: A Prospective Cohort Study
Brief Title: Oral Status as Predictors of Stroke-Associated Pneumonia and Swallowing Recovery in Patients With Post-Stroke Dysphagia
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0250
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Dsyphagia After Stroke
Keywords: Stroke; Deglutition; Dysphagia; Oral care; Swallowing disorder
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute stroke with dysphagia: Acute stroke patients with dysphagia

SUMMARY:
Post-stroke dysphagia (PSD) is a common condition that significantly impacts recovery and increases the risk of complications such as pneumonia, malnutrition, and prolonged hospital stays. Early identification and management are essential, as emphasized in several international clinical guidelines. However, predicting which patients will develop stroke-associated pneumonia (SAP) or experience delayed swallowing recovery remains a challenge. Recent evidence suggests that oral health status-including hygiene, tongue strength, and dental support-may play a key role in these outcomes. Assessing oral health could therefore aid in identifying high-risk patients and improving rehabilitation strategies.

Study Design and Setting A cohort study was designed with prospective data collection, conducted in parallel with a randomized controlled trial (RCT) at the stroke unit of Ghent University Hospital, Ghent, Belgium (ONZ-2024-0245). Data collection is expected to occur over two years, from 2025 to 2027.

The RCT is a one-day experimental study investigating the immediate effects of oral hygiene care on swallowing and masticatory functions. The interventions performed in this clinical study involve routine oral care procedures and are not expected to influence the outcomes of the cohort study.

Participants Participants will be recruited from all consecutive patients admitted to the stroke unit at Ghent University Hospital with ischemic or hemorrhagic stroke and a diagnosis of oropharyngeal dysphagia. For the diagnosis of oropharyngeal dysphagia, all patients will be restricted from oral intake upon arrival until a stroke nurse completes a step-by-step standardized protocol to screen for swallowing disorders.

DETAILED DESCRIPTION:
Data Collection A team of trained dental professionals and speech therapists will collect demographic and clinical data within the first three days after admission and will monitor cohort outcomes at day seven post-admission and weekly thereafter until discharge.

During the initial visit, baseline characteristics-including socio-demographic, medical, and clinical information-will be documented, with a specific focus on oral health status. Socio-demographic data will include age, gender, education level, living situation, and eligibility for increased healthcare cost reimbursement. Medical history will include smoking status, body mass index (BMI), medication use, stroke type, stroke location, and prior stroke events. Standardized assessment scores-namely the National Institutes of Health Stroke Scale (NIHSS), the Modified Rankin Scale (mRS), and the Functional Oral Intake Scale (FOIS)-will also be recorded. These data will be obtained from medical records and patient interviews conducted by the research team.

Oral status assessment includes two main components: dental information, and oral and masticatory function. Dental data will be gathered by a dentist using a standard dental probe, mirror, and headlamp at the bedside. Documented parameters will include oral care capacity, oral hygiene indices (dental plaque using a modified Turesky-Quigley-Hein index, tongue plaque via Winkel's index, and denture plaque assessed with the Augsburger and Elahi index). Additionally, oral disease status will be evaluated by measuring periodontal condition (Dutch Periodontal Screening Index - DPSI), tooth mobility (Miller's classification), clinical caries (International Caries Detection and Assessment System - ICDAS), and denture stomatitis (Newton's classification). Further oral status indicators will include the number of functional teeth, the number of posterior occluding pairs, denture status, and clinical signs of oral dryness.

Oral and masticatory function will be assessed using the Test of Masticating and Swallowing Solids (TOMASS), which evaluates the number of masticatory cycles, swallows, total time, and discrete bites while consuming a standardized cracker. Tongue strength will be measured using the Iowa Oral Performance Instrument during both resting and swallowing phases. Residual oral content will be scored using the Oral Residue Score-a 4-point scale (0-3) across eight oral regions: left teeth, right teeth, left sulcus and cheek, right sulcus and cheek, hard palate, soft palate, tongue dorsum, and floor of the mouth-yielding a maximum score of 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the stroke unit at Ghent University Hospital with ischemic or hemorrhagic stroke who are diagnosed with oropharyngeal dysphagia.
* Patients over 18 years of age with sufficient cognitive abilities and language skills to understand the swallowing exercises.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients with dysphagia
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pneumonia | At seven days post-admission and every seven days until discharge from the hospital or up to three months, whichever comes first.
  Diagnosed based on the modified Centers for Disease Control and Prevention criteria (Smith CJ, Kishore AK, Vail A, Chamorro A, Garau J, Hopkins SJ, et al. Diagnosis of stroke-associated pneumonia. Stroke. 2015)

SECONDARY OUTCOMES:
Oral intake status | At seven days post-admission and every seven days until discharge from the hospital or up to three months, whichever comes first.
  Oral intake status is interpreted for swallowing recovery and recorded as dichotomous data, with recovered swallowing defined as FOIS (Functional Oral Intake Scale) greater than five and unrecovered swallowing as FOIS equal to or less than five.
Length of hospital stays | At seven days post-admission and every seven days until discharge from the hospital or up to three months, whichever comes first.
  Length of Stay refers to the total duration of time a patient spends in a hospital
In-hospital mortality | At seven days post-admission and every seven days until discharge from the hospital or up to three months, whichever comes first.
  Death occurring during the hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
The IPD must be shared as anonymized or pseudonymized information, which may be included in a meta-analysis upon request. Data transfer must be conducted under Ghent University Hospital conditions, with legal experts drafting and reviewing the agreement (https://hiruz.be/cu/). Additionally, any data containing personal information requires approval from the Ethics Committee before transfer.